CLINICAL TRIAL: NCT01183494
Title: A Genotype-guided Phase I Study of Irinotecan Administered in Combination With 5-fluorouracil/Leucovorin (FOLFIRI) and Bevacizumab in Advanced Colorectal Cancer Patients
Brief Title: A Genotype-guided Study of Irinotecan Administered in Combination With 5-fluorouracil/Leucovorin (FOLFIRI) and Bevacizumab in Advanced Colorectal Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-277-B
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UGT1A1*1/*1 (Experimental): Participants with UGT1A1*/*1 genotype will receive escalating doses of FOLFIRI (folinic acid+fluorouracil+irinotecan) and bevacizumab. The initial dose of irinotecan will be 260 mg/m2 administered as a 120 min intravenous infusion every two weeks. The dosage of irinotecan will be increased to 310, 370, and 420 mg/m2, and further irinotecan doses will be increased by 14%. 5-FU will be administered as a 400 mg/m2 bolus right after the end of the irinotecan infusion, followed by 2,400 mg/m2 over a 46 h continuous infusion plus LV 200 mg/m2 every two weeks. Bevacizumab will be administered at a dose of 5 mg/kg over 15-30 min IV (after an initial 90 min infusion without a reaction) every two weeks. The first dose will be administrated on day 2 (48 hours after the first irinotecan administration), while the second dose on day 14 (the same day as the second irinotecan administration). No dose escalation will be performed for 5-FU, LV or bevacizumab.
  Interventions: Drug: FOLFIRI, Avastin, Irinotecan
- UGT1A1*1/*28 (Experimental): Participants with UGT1A1*1/*28 genotype will receive escalating doses of FOLFIRI (folinic acid+fluorouracil+irinotecan) and bevacizumab. The initial dose of irinotecan will be 260 mg/m2 administered as a 120 min intravenous infusion every two weeks. The dosage of irinotecan will be increased to 310, 370, and 420 mg/m2, and further irinotecan doses will be increased by 14%. 5-FU will be administered as a 400 mg/m2 bolus right after the end of the irinotecan infusion, followed by 2,400 mg/m2 over a 46 h continuous infusion plus LV 200 mg/m2 every two weeks. Bevacizumab will be administered at a dose of 5 mg/kg over 15-30 min IV (after an initial 90 min infusion without a reaction) every two weeks. The first dose will be administrated on day 2 (48 hours after the first irinotecan administration), while the second dose on day 14 (the same day as the second irinotecan administration). No dose escalation will be performed for 5-FU, LV or bevacizumab.
  Interventions: Drug: FOLFIRI, Avastin, Irinotecan

INTERVENTIONS:
Drug: FOLFIRI, Avastin, Irinotecan — Patients will be treated with the FOLFIRI regimen plus bevacizumab. Irinotecan will be administered at doses higher than the standard dose in patients with the UGT1A1*1/*1 and UGT1A1*1/*28 genotypes, while the doses of infusional 5-FU/LV and bevacizumab will remain unchanged.

SUMMARY:
This study is being done to determine the maximum dose of a certain chemotherapy drug (irinotecan) that can be tolerated as part of a combination of drugs. There is a combination of chemotherapy drugs typically used to treat cancer of the colon and rectum: 5-Flurouracil (5-FU), leucovorin, and irinotecan; the combination is known as FOLFIRI. At the present time, the Food and Drug Administration (FDA) has approved this drug combination for the treatment of cancers of the colon and rectum. The FDA has also approved the use of a drug called bevacizumab (or Avastin) in combination with FOLFIRI, and this is considered one of the standards of care for all patients with colon and rectal cancer which has spread.

The best dose of irinotecan to use in the combination of FOLFIRI and bevacizumab is not known. Earlier studies have shown that higher doses of irinotecan can be used safely as part of the FOLFIRI combination, but it is unclear whether these same doses will be safe when bevacizumab is added to this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of metastatic colorectal adenocarcinoma
2. No prior chemotherapy for metastatic disease
3. Age ≥18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (5. Life expectancy > 3 months
5. Adequate organ function, including bone marrow (absolute neutrophil count (ANC) ≥l500/μl, haemoglobin ≥ 9g/dL, platelets ≥ 100,000/ μl); hepatic (total bilirubin < 1.6 mg/dl;SGOT and SGPT < 2.5 x upper limit of normal for patients without liver metastases and < 5x upper limit of normal for patients with liver metastases); and renal (serum creatinine ≤ 1.5x upper limit of normal).
6. Patients who are eligible to be registered in the study, based upon the above criteria, will be genotyped for the UGT1A1*28 polymorphism and stratified into two groups based on the presence of the UGT1A1*1/*1 or UGT1A1*1/*28 genotype.
7. Patients with the UGT1A1*28/*28 genotype or carriers of the other alleles (TA5 and TA8)will be excluded.
8. For patients to be evaluable for response (a secondary end point), they must have at least one measurable lesion as defined by RECIST (i.e., lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral CT scan).
9. Patients without measurable lesions can be included and will be evaluated only for toxicity.
10. Signed informed consent and local IRB approval is required.
11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, up until 30 days after final study treatment. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Prior irinotecan or bevacizumab treatment
2. Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
3. Diarrhea greater than grade 1
4. Bowel obstruction
5. Documented brain metastases
6. Serious active infectious disease
7. Active uncontrolled bleeding or fistulas
8. Pregnancy
9. Radiotherapy or major surgery within 4 weeks
10. Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been disease-free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12-12 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 years
  To define the Maximum Tolerated Dose (MTD), the Dose Limiting Toxicity (DLT), and the recommended dosage of irinotecan administered in first-line therapy with FOLFIRI plus bevacizumab for patients with metastatic CRC and either the UGT1A1*1/*1 or UGT1A1*1/*28 genotype.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of irinotecan in combination with bevacizumab. | 3 years
  To evaluate the effect of bevacizumab on the pharmacokinetics of irinotecan.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, MD, Principal Investigator — University of Chicago
Locations (2):
- The University of Chicago, Chicago, Illinois, United States
- CRO-National Cancer Institute, Aviano, Italy